CLINICAL TRIAL: NCT04843657
Title: Objective Data for Cancer Related Fatigue in Cancer Patients
Brief Title: Precise Care for Cancer Related Fatigue
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: cancer related fatigue monitor
Record Dates: First submitted 2021-04-12; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Cancer-Related Condition
Keywords: Cancer-related fatigue; smart bracelet device; symptoms for subjective and objective
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microbiota
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Observation for symptom distress — Observation for symptom distress

SUMMARY:
This project expects to enroll 200 cancer patients and their subjective-objective measurements on fatigue, stress, symptoms, and total steps will be validated so that the information can be used in further care and improvement of life of quality of the patients.

ELIGIBILITY:
Inclusion Criteria:

- Age ≧ 20 years old; One group had a cancer diagnosis, one group no cancer diagnosis; Can continuous wearing bracelet for 7 days or more

Exclusion Criteria:

- Unclear and unable to answer the questionnaire

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with some cancer treatment side effects.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
fatigue | 7-8 days
  severity of fatigue level; measurement tool: Brief Fatigue Index
Heart Rate Variability (HRV) monitor | 7-8 days
  Use a digital device to measure the heart rate variability and calculate the HRV data

SECONDARY OUTCOMES:
Distress Thermometer(DT) | 7-8 days
  a screening measure to identify and address psychological distress in individuals with cancer. a cutoff score of 3 on the DT to indicate patients with clinically elevated levels of distress.
Leeds Sleep Evaluation Questionnaire(LSEQ） | 7-8 days
  To assess sleep quality, higher scores mean more disrupt sleep.
International Physical Activity Questionnaire(IPAQ） | 7-8 days
  Life activity survey
Perceived Stress Scale (PSS） | 7-8 days
  higher scores mean more stressful condition
ESAS (Edmonton Symptom Assessment Scale) | 7-8 days
  higher scores mean more severe symptoms condition

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Wei Huang, Principal Investigator — Taipei Medical University

IPD SHARING:
Plan to Share IPD: Undecided